CLINICAL TRIAL: NCT01956799
Title: Identification of Mechanisms in the Erythroid Response in Patients With Myelodysplasia Undergoing Chelation Therapy
Brief Title: Identification of Mechanism in the Erythroid Response in Patients With Myelodysplasia Undergoing Chelation Therapy
Acronym: BIOFER12
Status: Completed | Type: Observational
Sponsor: Fondazione Italiana Sindromi Mielodisplastiche-ETS (Other)
Responsible Party: Sponsor
Other Study IDs: FISM-BIOFER12
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Myelodysplasia; Myelofibrosis; Aplastic Anemia
Keywords: MDS; PMF; CMML; AA
MeSH Terms: conditions — Anemia, Refractory, with Excess of Blasts; Primary Myelofibrosis; Anemia, Aplastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood and bone marrow
Oversight: Data Monitoring Committee: No

SUMMARY:
The study aims to evaluate the molecular mechanism underlying the erythroid response observed in some patients with myelodysplasia, myelofibrosis and aplastic anemia treated with Deferasirox or Deferoxamina.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 and older
2. Diagnosis of Myelodysplasia, myelofibrosis or aplastic anemia
3. transfusion-dependent anemia undergoing chelation therapy with deferasirox or deferoxamine

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of Myelodysplasia, myelofibrosis or aplastic anemia undergoing chelation therapy with deferasirox or deferoxamine
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2018-07 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
To assess the molecular mechanism underlying the erythroid response | 12 months
  The primary outcome is to evaluate the molecular mechanism underlying the erythroid response (hemogoblin increase and reduction or elimination of trasfusion dependence) observed in some patients with myelodysplasia, myelofibrosis and aplastic anemia treated with Deferasirox or Deferoxamina

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Cilloni, MD, Principal Investigator — AOU S. Luigi Gonzaga, Regione Gonzole 10, 10043 Orbassano (TO)
Locations (20):
- Italy (20):
  - Ematologia, AO SS. Antonio e Biagio, Alessandria, AL
  - Clinica di Ematologia, AOU Ospedale di Torrette, Ancona, AN
  - Ematologia con trapianto, AOU Policlinico di Bari, Bari, BA
  - Istituto di Ematologia e Oncologia Medica, Policlinico S.Orsola, Bologna, BO
  - Ematologia, Spedali Civili, Brescia, BS
  - Struttura complessa di Ematologia, ASO S.Croce e Carle, Cuneo, CN
  - Cattedra di Ematologia Policlino Careggi, Florence, FI
  - Clinica Ematologica, Università di Genova, Genova, GE
  - U.O. Clinica Medicina Interna, IRCCS San Martino IST, Genova, GE
  - UO Ematologia e CTMO, Ospedale Civile G. da Saliceto, Piacenza, PC
  - Ematologia, Università di Padova, Padua, PD
  - Struttura Cattedra di Ematologia e CTMO, AOU di Parma, Parma, PR
  - Ematologia e Centro Trapianti, Centro di Riferimento Oncologico della Basilicata, Rionero in Vulture, PZ
  - Medicina Interna II Divisione di Ematologia, Ospedale S. Luigi Gonzaga, Orbassano, TO
  - Ematologia 2, AOU Città della Salute e della Scienza, Torino, TO
  - S.C.D.U. Ematologia e Terapie cellulari, Ospedale Mauriziano, Torino, TO
  - UOC Ematologia, Ospedale S.Eugenio, Roma
  - Policlinico A.Gemelli, Roma
  - UOC Ematologia, AO S. Giovanni Addolorata, Roma
  - Ematologia, AO S. Andrea, Roma